CLINICAL TRIAL: NCT00912639
Title: A Clinical Trial of Paclitaxel Loaded Polymeric Micelle (Genexol-PM®) in Patients With Taxane-Pretreated Recurrent Breast Cancer
Brief Title: A Clinical Trial of Paclitaxel Loaded Polymeric Micelle in Patients With Taxane-Pretreated Recurrent Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Korean Breast Cancer Study Group (Other)
Responsible Party: Byung-Joo Song, The Catholoic university of Korea, St. Mary's hospital.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KBCSG004
Record Dates: First submitted 2009-05-31; First posted 2009-06-03 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Recurrent Breast Cancer
Keywords: recurrent breast cancer; Genexol-PM
MeSH Terms: conditions — Breast Neoplasms | interventions — genexol-PM

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Genexol-PM (Experimental): All the patients are recurrent breast cancer after taxane treatment. Patients with a measurable lesion (at least 1 measurable lesion)
  1. Spiral CT : lesion ≥ 10mm (unidimension)
  2. X-ray, MRI, ultrasound : lesion ≥ 20 mm (unidimension)
  Interventions: Drug: Paclitaxel loaded Polymeric micelle

INTERVENTIONS:
Drug: Paclitaxel loaded Polymeric micelle — Genexol-PM at a dose of 300mg/m2 was diluted in 500 ml of 5% dextrose solution or normal saline and infused i.v. for 3 h on day 1.Treatment was repeated every 3 weeks until either disease progression or intolerance. A minimum of 6 cycles was recommended.
  Other Names: Genexol-PM®

SUMMARY:
The purpose of this study is to evaluate the response rate in patients with taxane-pretreated recurrent breast cancer receiving paclitaxel loaded polymeric micelle (Genexol-PM).

DETAILED DESCRIPTION:
Genexol-PM is a novel Cremophor EL-free polymeric micelle formulation of paclitaxel. This single arm, multicenter phase IV study was designed to evaluate the response rate, toxicity, progression free survival and tumor control rate of Genexol-PM in patients with Taxane-pretreated recurrence breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged >=18 years
2. WHO (ECOG) performance status 0-2
3. Estimated life expectancy of >=3 months
4. Have given written informed consent and are available for prolonged follow-up

Exclusion Criteria:

1. Patients with previous chemotherapy for recurrent breast cancer
2. Breast cancer recurrence within 12 months after taxane treatment
3. Her-2/neu expression
4. Patients with malignancies (other than breast cancer) within the last 5 years, except for adequately treated in situ carcinoma of the cervix or basal cell, squamous cell carcinoma of the skin.
5. Brain metastasis
6. uncontrolled infection, medically uncontrollable heart disease
7. other serious medical illness or prior malignancies
8. Pregnant or lactating women were excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Response rate was assessed by imaging using the RECIST (Response Evaluation Criteria In Solid Tumor) guideline | 1 year

SECONDARY OUTCOMES:
Toxicity | 1 year
Progression Free Survival | 1 year
Tumor control rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Joo Song, MD.PhD., Principal Investigator — The Catholoic university of Korea, St. Mary's hospital.
Locations (1):
- Department of surgery, The Catholoic university of Korea, St. Mary's hospital., Seoul, South Korea